CLINICAL TRIAL: NCT03393780
Title: Prospective Multicentre Non-Interventional Study to Assess the Patterns of Use of REKOVELLE® in Women Undergoing In Vitro Fertilisation or Intracytoplasmic Sperm Injection Procedures in Routine Clinical Practice
Brief Title: Study to Assess the Patterns of Use of REKOVELLE® in Naïve Women Undergoing In Vitro Fertilisation or Intracytoplasmic Sperm Injection Procedures
Acronym: PROFILE
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000300
Record Dates: First submitted 2017-12-13; First posted 2018-01-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2020-11

CONDITIONS: Controlled Ovarian Stimulation
MeSH Terms: interventions — follitropin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Follitropin Delta — The Intervention (solution for injection) is delivered with an injection pen. The REKOVELLE® dose will be based on recent determination (within the last 12 months) of AMH (anti- müllerian hormone) measured by the following diagnostic test from ROCHE: ELECSYS AMH Plus immunoassay.
  Other Names: REKOVELLE®

SUMMARY:
The purpose of this study is to monitor the use in routine clinical practice of REKOVELLE®. This study will collect information from patients who never underwent previous in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) treatments for up to three consecutive treatment cycles.

The ovarian stimulation protocol with REKOVELLE®, a new recombinant human Follicle Stimulating Hormone (FSH) prescribed for ovarian stimulation, is individualised with a dosing regimen that is based on two parameters: the body weight and the level of a hormone, the Anti Müllerian Hormone, (AMH), a parameter used to predict how the ovaries will respond to the ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria: Patients who meet all of the following criteria are eligible for participation:

* Females are prescribed REKOVELLE® for their first in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) treatment cycle using fresh or frozen ejaculated sperm from male partner or sperm donor
* Willing and able to provide written informed consent

Exclusion Criteria: Patients who meet any of the following criteria are not eligible for participation:

* Participating in an interventional clinical trial in which any treatment or follow-up is mandated
* Women with a contraindication for prescription of REKOVELLE® treatment
* Oocyte donors
* Women undergoing ovarian stimulation for fertility preservation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who are prescribed REKOVELLE® within the approved indication for IVF or ICSI for their first in vitro fertilisation treatment will be invited to participate in the study. Patients will be enrolled only after the treatment decision has been made and no aspect of this study will interfere with or influence the routine medical procedures and/or medications received
Sampling Method: Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Use of algorithm-based individualised dosing regimen to decide daily dose of REKOVELLE® | At consultation visit where the daily dose of REKOVELLE® is decided
  Calculated with body weight in kilograms or pounds and AMH serum level in pmoL/L or ng/ml to define the daily dose of REKOVELLE® in micrograms
Use of the dosing App | At consultation visit where the daily dose of REKOVELLE® is decided
  Use of the Ferring developed dosing app for the daily dose calculation by answering yes/no to a questionnaire
Daily dose of REKOVELLE® in micrograms | From day 1 up to day 20 of REKOVELLE® stimulation
Number of days of treatment with REKOVELLE® | From day 1 up to day 20 of REKOVELLE® stimulation
  Adjusted during the stimulation based on blood sample of Oestrogen levels and number of follicles (at the discretion of the investigator)
Day of REKOVELLE® stimulation start | At the day of the first REKOVELLE® injection during the ovarian stimulation treatment
  The time point of the start of the stimulation is decided at the discretion of the investigator
Day of REKOVELLE® stimulation end | At the day of the last REKOVELLE® injection during the ovarian stimulation treatment
  The time point of the end of the stimulation is decided at the discretion of the investigator
Type of GnRH used for Lutenizing Hormone(LH) surge suppression | At consultation visit where the LH surge suppression protocol is decided
  Defined as a choice between GnRH agonist and GnRH antagonist
Day of LH surge suppression protocol start | At the day of the first GnRH administration during the ovarian stimulation treatment
  The time point of the start of LH surge suppression is decided at the discretion of the investigator
Day of LH surge suppression protocol end | At the day of the last GnRH administration during the ovarian stimulation treatment
  The time point of the end of LH surge suppression is decided at the discretion of the investigator
Type of drug used for the triggering of follicle maturation | At consultation visit where the triggering of follicle maturation protocol is decided
  Decided as a choice between hCG and/or GnRH
Date of administration of hCG and/or GnRH for follicle maturation | At the day of administration (at the discretion of the investigator)
  Date when the investigator decides to trigger the final follicle maturation
Type of drug used for Luteal phase support | From ovum pick-up day (the length of luteal phase support is decided at the discretion of the investigator)
  Decided as a choice between Progesterone, Oestrogen and hCG
Parameters used to define the daily dose of REKOVELLE® in case a new assisted reproductive technology treatment is initiated | At consultation visit where the ovarian stimulation treatment strategy is decided
  According to the Summary of Product Characteristics, the daily dose can be increased or decreased for subsequent cycles based on the patient response to the initial treatment cycle.

CONTACTS AND LOCATIONS:
Locations (10):
- Melbourne - IVF (there may be other sites in this country), East Melbourne, Australia
- Landeskrankenhaus Feldkirch Kinderwunschzentrum (there may be other sites in this country), Feldkirch, Austria
- UZ Brussel (there may be other sites in this country), Brussels, Belgium
- Clinique - OVO (there may be other sites in this country), Montreal, Canada
- Viva Neo Praxisklinik Sydow (there may be other sites in this country), Berlin, Germany
- Policlinico di Milano (there may be other sites in this country), Milan, Italy
- Erasmus Medisch Centrum (there may be other sites in this country), Rotterdam, Netherlands
- Invicta Fertility Clinic Gdansk (there may be other sites in this country), Gdansk, Poland
- Clinica Eugin (there may be other sites in this country), Barcelona, Spain
- The London Women Clinic (there may be other sites in this country), London, United Kingdom

REFERENCES:
- [Result] Blockeel C, Griesinger G, Rago R, Larsson P, Sonderegger YLY, Riviere S, Laven JSE. Prospective multicenter non-interventional real-world study to assess the patterns of use, effectiveness and safety of follitropin delta in routine clinical practice (the PROFILE study). Front Endocrinol (Lausanne). 2022 Dec 22;13:992677. doi: 10.3389/fendo.2022.992677. eCollection 2022. PMID 36619578